CLINICAL TRIAL: NCT01484613
Title: Effectiveness and Reliability of Selected Site Pacing for Avoidance of Phrenic Nerve Stimulation in CRT Patients With Quadripolar LV Leads
Brief Title: Selected Site Pacing to Avoid Phrenic Nerve Stimulation in Cardiac Resynchronization Patients With Quadripolar Left Ventricular Leads
Acronym: EffaceQ
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: H56
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Hear Failure; Cardiac resynchronization; CRT-D; quadripolar
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quadripolar lead: All participants receive a CRT-D system with quadripolar lead
  Interventions: Device: quadripolar LV lead (Quartet)

INTERVENTIONS:
Device: quadripolar LV lead (Quartet) — All participants will receive CRT-D system with a quadripolar lead. This lead offers 10 LV lead vectors to choose from
  Other Names: Quartet

SUMMARY:
Cardiac resynchronization (CRT) therapy is well established for treatment of patients with severe heartfailure, reduced left ventricular (LV) function and ventricular dyssynchrony. Roughly 1/3 of CRT patients do not improve after CRT implant. One possible reason is interruption of biventricular pacing. This might be caused by several conditions, including elevated left ventricular (LV) pacing thresholds or presence of phrenic nerve stimulation (PNS). CRT devices with quadripolar LV leads offer 10 LV pacing vectors to choose from. It's the aim of this prospective observational study to investigate efficacy and reliability of cardiac resynchronization therapy (CRT) with quadripolar left ventricular leads.

Hypothesis: In more than 90% of patients, who received a CRT system with quadripolar LV lead, at least one acceptable LV lead vector is available.

DETAILED DESCRIPTION:
Definition of an acceptable lead vector: Any LV pacing vector that complies in both tested body positions (left lateral position and sitting) with both criteria:

1. Phrenic nerve stimulation threshold is at least twice as high as LV pacing threshold
2. LV pacing threshold is less or equals 2.5Volts (V) @0.5 milliseconds (ms)

ELIGIBILITY:
Inclusion Criteria:

* Indication for implantation of a CRT-D
* Age >= 18 years
* Written informed consent

Exclusion Criteria:

* Already implanted LV or coronary sinus lead
* Previous unsuccessful LV lead implant attempt
* Patient is eligible for heart transplantation
* Comorbidities that results in life expectancy of less than 12 months
* Known pregnancy
* Inability to provide written patient informed consent
* Participation to another study with active treatment arm (i.e. randomized studies etc...)
* Patient is not willing or is not able to visit the study center for the study assessments within the first 3 months after implant
* Patient is not able to understand or answer the quality of life questionaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are planned for being implanted with a cardiac resynchronization therapy implantable cardioverter defibrillator (CRT-D) system in the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least one acceptable lead vector | Pre hospital discharge (PHD) to 3 months
  Definition of acceptable lead vector:
  Any LV vector that complies in both tested body positions with both criteria:
  1. Phrenic nerve stimulation threshold is at least twice as high as LV pacing threshold
  2. LV pacing threshold is less or equals 2.5V@0.5ms

SECONDARY OUTCOMES:
Quality of Life | Baseline to 3 months
  Minnesota living with heart failure questionaire
Phrenic nerve stimulation (PNS) | PHD to 3 months
  * Incidence of PNS per LV pacing vector
  * Freedom from PNS for the permanently programmed LV vector
LV pacing thresholds | PHD to 3 months
  * LV pacing thresholds per LV vector
  * Incidence of elevated (>2.5V/0.5ms) LV pacing thresholds per LV vector
Number of acceptable LV lead vectors per patient | PHD to 3 months
Finally programmed LV lead vector | PHD to 3 months
  * Need for reprogramming
  * Percentage of patients with conventional (bipolar) and extended (quadripolar) LV vectors

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Brachmann, Prof., Principal Investigator — Klinikum Coburg GmbH
Locations (16):
- Germany (16):
  - Klinikum Coburg GmbH, Coburg
  - Evangelisches Krankenhaus Kalk, Cologne
  - Krankenhaus Mörsenbroich-Rath GmbH, Düsseldorf
  - Klinikum Esslingen, Esslingen am Neckar
  - Cardioangiologisches Centrum Bethanien, Frankfurt am Main
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Herz- und Gefäßzentrum am Krankenhaus Neu-Bethlehem, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - St.-Marien-Hospital GmbH, Lünen
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Marien-Hospital, Marl
  - Klinikum Großhadern der Ludwig-Maximilians-Universität München, München
  - Universitätsklinikum Münster, Münster
  - Niels-Stensen-Kliniken Marienhospital Osnabrück, Osnabrück
  - Klinikum Dorothea Christiane Erxleben GmbH, Quedlinburg